CLINICAL TRIAL: NCT00948051
Title: A Placebo-controlled, Double-blind Randomized Study to Evaluate the Efficacy of a follow-on Milk Formula Supplemented With Fructo-oligosaccharides on Immune Response in Healthy Infants
Brief Title: Effects of follow-on Formula Enriched on Short-chain Fructooligosaccharides (scFOS) on Immune Response in Healthy Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syral (Industry)
Responsible Party: Frederique Respondek/ Scientific Affairs Manager, Syral
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: FOS_FOF08
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Infant
MeSH Terms: interventions — fructooligosaccharide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Fructo-oligosaccharides (Experimental)
  Interventions: Dietary Supplement: Follow-on formula supplemented with fructo-oligosaccharides
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Follow-on formula enriched with placebo (maltodextrins)

INTERVENTIONS:
Dietary Supplement: Follow-on formula supplemented with fructo-oligosaccharides — Follow-on formula supplemented with fructo-oligosaccharides
  Arms: Fructo-oligosaccharides
Dietary Supplement: Follow-on formula enriched with placebo (maltodextrins) — Follow-on formula enriched with placebo (maltodextrins)
  Arms: Placebo

SUMMARY:
In this study the investigators hypothesized that the chronic intake of fructo-oligosaccharides would increase fecal immunoglobulin A (IgA) specific to poliovirus vaccination and bifidobacteria in infants.

ELIGIBILITY:
Inclusion Criteria:

* infants aged of 4 months at randomization
* not breast-fed infants

Exclusion Criteria:

* infants suffering from a chronic or severe disease susceptible to interfere with one of the evaluation criteria
* infants suffering from a disease associated with gastro-intestinal disorder
* infants who have taken antibiotic during the 2 months preceding randomization

Ages: 4 Months to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of the intake of a follow-on milk formula supplemented with FOS in increasing infant's response to vaccination | 1 month

SECONDARY OUTCOMES:
To evaluate the impact of the intake of a follow-on milk formula supplemented with FOS in increasing infant's faecal bifidobacteria concentration | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Tormo, Barcelona, Spain